CLINICAL TRIAL: NCT00488488
Title: A Non-Interventional Study To Evaluate The Safety And Effectiveness Of Tygacil In The Treatment Of Patients With Complicated Intra-Abdominal Infections Or Complicated Skin And Skin Structure Infections
Brief Title: A Pharmacovigilance Evaluation And Assessment Of The Prescribing Practice For Tygacil In Usual Health Care Setting
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Other Study IDs: 3074A1-102045; B1811054 (Other: Pfizer)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2011-07-18 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-06

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: tigecycline

INTERVENTIONS:
Drug: tigecycline — The patients will be treated in accordance with the requirements of the labeling of tigecycline in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: Tygacil

SUMMARY:
To assess the efficacy and safety of Tygacil in the usual German hospital setting. The main goals are: to assess the efficacy of Tygacil under usual care conditions (cure rate); to assess the main side effects observed in daily medical practice (Safety of Tygacil); to determine whether patients are optimally dosed with Tygacil (according to the label) and the proportion of patients receiving a monotherapy versus combination therapy; to observe the potential resistance development against Tygacil in Germany; to determine which antibiotic agents are chosen for a combination therapy with Tygacil; to determine to which antibiotic substance non-responders to Tygacil are switched; to assess the duration of the intravenous therapy with Tygacil and to determine whether and which patients receive an oral antibiotic substance after the therapy with Tygacil; to collect information on profile, comorbidities and characteristics of patients treated with Tygacil.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician.

ELIGIBILITY:
Inclusion Criteria:

* Actual or planned therapy with tigecycline.
* At least 18 years old.

Exclusion Criteria:

* Hypersensitivity to antibiotics or tigecycline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (i.e., at least 18 years old) with a verified diagnosis of complicated Intra-Abdominal Infection (cIAI) or complicated Skin and Skin Structure Infection (cSSSI), for whom the decision for Tygacil treatment had already been made.
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Bassetti M, Eckmann C, Bodmann KF, Dupont H, Heizmann WR, Montravers P, Guirao X, Capparella MR, Simoneau D, Sanchez Garcia M. Prescription behaviours for tigecycline in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii5-14. doi: 10.1093/jac/dkt140. PMID 23772047
- [Derived] Guirao X, Sanchez Garcia M, Bassetti M, Bodmann KF, Dupont H, Montravers P, Heizmann WR, Capparella MR, Simoneau D, Eckmann C. Safety and tolerability of tigecycline for the treatment of complicated skin and soft-tissue and intra-abdominal infections: an analysis based on five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii37-44. doi: 10.1093/jac/dkt143. PMID 23772045
- [Derived] Montravers P, Bassetti M, Dupont H, Eckmann C, Heizmann WR, Guirao X, Garcia MS, Capparella MR, Simoneau D, Bodmann KF. Efficacy of tigecycline for the treatment of complicated skin and soft-tissue infections in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii15-24. doi: 10.1093/jac/dkt141. PMID 23772042
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074A1-102045&StudyName=A%20Pharmacovigilance%20Evaluation%20And%20Assessment%20Of%20The%20Prescribing%20Practice%20For%20Tygacil%20In%20Usual%20Health%20Care%20Setting

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional study; participants were selected and treated according to the usual clinical practice of their physician.
Pre-assignment Details: A total of 1,028 participants were documented at 137 observational sites. Three participants were excluded from analysis due to retrospective documentation.
Groups:
- Tygacil: Tygacil prescribed according to product label; recommended dose 100 milligrams (mg) initial dose, then 50 mg every 12 hours; maximum dose 100 mg per day
Period: Overall Study
Arm/Group | Tygacil
Started | 1028
Analyzed | 1025 (3 participants were not analyzed due to retrospective documentation.)
Completed | 760 (Excludes 4 participants with missing information.)
Not Completed | 268

BASELINE CHARACTERISTICS:
Arm/Group | Tygacil
Number analyzed (Participants) | 1025
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (13.7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 380
  Male | 642
  Missing Data (Unspecified) | 3
Resistance Patterns at Baseline: Percentage of Participants with Resistant Pathogens [Number; unit: percentage of participants] — Participants with baseline pathogen data documented that had pathogens found to be resistant; n = number of participants with specified pathogen.
  percentage of participants
    Pseudomonas aeruginosa (n=23) | 73.9
    Proteus vulgaris (n=3) | 33.3
    Proteus mirabilis (n=6) | 16.7
    Other pathogens (unspecified) (n=30) | 13.3
    Enterobacter species (spp) (n=26) | 3.8
    Klebsiella pneumoniae (n=29) | 3.4
    Enterococcus faecalis (n=65) | 1.5
    Escherichia coli (n=99) | 1.0
    Enterococcus faecium (n=146) | 0
    Staphylococcus aureus (n=120) | 0
    Staphylococcus spp (n=63) | 0
    Klebsiella oxytoca (n=16) | 0
    Stenotrophomonas maltophilia (n=8) | 0
    Streptococcus pyogenes (A group) (n=7) | 0
    Other clostridiae (n=6) | 0
    Citrobacter freundii (n=5) | 0
    Streptococcus anginosus group (n=5) | 0
    Other Bacteroides species (n=5) | 0
    Acinetobacter spp. (n=4) | 0
    Bacteroides fragilis (n=3) | 0
    Haemophilus spp (n=2) | 0
    Streptococcus pneumoniae (n=2) | 0
    Peptostreptococcus (n=2) | 0
    Serratia spp (n=1) | 0
    Morganella morganii (n=1) | 0
    Bacteroides thetaiotamicron (n=1) | 0
    Streptococcus agalactiae (B group) (n=1) | 0
    Clostridium perfringens (n=1) | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical and Microbiological Cure: All Participants
Description: Cure = complete resolution of infection symptoms; no further antibiotic treatment required. A second microbiological examination was documented only for participants with treatment failure.
Time Frame: End of Treatment (duration based on severity, location, and clinical response; maximum duration 47 days)
Population: All participants: participants exposed to Tygacil who had non-retrospective post-baseline data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 1025
percentage of participants | 33.8 [30.9 to 36.7]

2. Primary Outcome: Percentage of Participants With Clinical and Microbiological Cure: Nosocomial Infections
Description: as for outcome 1
Time Frame: End of Treatment (duration based on severity, location, and clinical response; maximum duration 47 days)
Population: All participants; N = number of participants with nosocomial infections.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 658
percentage of participants | 29.0 [25.6 to 32.7]

3. Primary Outcome: Percentage of Participants With Clinical and Microbiological Cure: Community-acquired Infections
Description: as for outcome 1
Time Frame: End of Treatment (duration based on severity, location, and clinical response: maximum duration 47 days)
Population: All participants; N = number of participants with community-acquired infections.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 344
percentage of participants | 43.9 [38.6 to 49.3]

4. Primary Outcome: Percentage of Participants With Composite Cure: All Participants
Description: Composite Cure = complete resolution or improvement of infection symptoms; no further antibiotic treatment required.
Time Frame: End of Treatment (duration based on severity, location, and clinical response; maximum duration 47 days)
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 1025
percentage of participants | 74.2

5. Primary Outcome: Percentage of Participants With Composite Cure: Nosocomial Infections
Description: Composite Cure = complete resolution or improvement of infection symptoms; no further antibiotic treatment required.
Time Frame: End of Treatment (duration based on severity, location, and clinical response; maximum duration 47 days)
Population: All participants; N = number of participants with nosocomial infections.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 658
percentage of participants | 70.5

6. Primary Outcome: Percentage of Participants With Composite Cure: Community-acquired Infections
Description: Composite Cure = complete resolution or improvement of infection symptoms; no further antibiotic treatment required.
Time Frame: End of Treatment (duration based on severity, location, and clinical response: maximum duration 47 days)
Population: All participants; N = number participants with community-acquired infections.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 344
percentage of participants | 82.3

7. Secondary Outcome: Participants With Probable Failure at Follow-up
Description: Participants with antibiogram follow-up due to treatment failure who had detectable pathogens. Treatment failure = no significant improvement of infection symptoms under Tygacil therapy.
Time Frame: Follow-up (up to Day 47)
Population: All participants.
Measure: Number; unit: participants
Arm/Group | Tygacil
Number analyzed (Participants) | 1025
participants | 162

8. Secondary Outcome: Percentage of Participants With Resistant Pathogens Identified at Follow-up Due to Treatment Failure
Description: Percentage of participants with resistant pathogens for each pathogen identified at second (follow-up) microbial examination. A second microbiological examination was documented only for participants with treatment failure. Treatment failure = no significant improvement of infection symptoms under Tygacil therapy.
Time Frame: Follow-up (up to Day 47)
Population: All participants; N = number of participants who had a follow-up microbial investigation due to treatment failure; n = number of participants who tested positive for pathogen and had isolates tested for pathogen resistance.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 162
percentage of participants
  Pseudomonas aeruginosa (n=12) | 100.0
  Other pathogens (unspecified) (n=6) | 100.0
  Klebsiella oxytoca (n=1) | 100.0
  Proteus mirabilis (n=6) | 50.0
  Proteus vulgaris (n=2) | 50.0
  Stenotrophomonas maltophilia (n=4) | 25.0
  Klebsiella pneumoniae (n=9) | 22.2
  Enterococcus faecalis (n=10) | 20.0
  Enterobacter species (spp) (n=11) | 18.2
  Escherichia coli (n=14) | 7.1
  Staphylococcus aureus (n=16) | 6.3
  Enterococcus faecium (n=15) | 0
  Staphylococcus spp (n=5) | 0
  Serratia spp (n=2) | 0
  Citrobacter freundii (n=1) | 0
  Acinetobacter spp. (n=1) | 0

9. Secondary Outcome: Antibiotic Agents Chosen for Combination Therapy With Tigecycline
Description: Percentage of participants who received each antibiotic administered as combination therapy with tigecycline.
Time Frame: Baseline to End of Treatment (up to Day 47)
Population: All participants; N = number of participants who were concomitantly treated with other antibiotics in combination with Tygacil; n = number of participants who were concomitantly treated with specified antibiotic in combination with Tygacil.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 512
percentage of participants
  ceftazidime (n=191) | 18.6
  ciprofloxacin (n=62) | 6.0
  fluconazole (n=59) | 5.8
  meropenem (n=49) | 4.8
  metronidazole (n=48) | 4.7
  vancomycin (n=27) | 2.6
  cefepime (n=26) | 2.5
  pip/tazo (n=18) | 1.8
  piperacillin (n=14) | 1.4
  caspofungin (n=13) | 1.3
  levofloxacin (n=13) | 1.3
  other antimycotics for system use (n=13) | 1.3
  imipenem (n=12) | 1.2
  primaxin (n=12) | 1.2
  voriconazole (n=11) | 1.1
  erythromycin (n=10) | 1.0
  gentamicin (n=10) | 1.0
  sulbactam (n=10) | 1.0
  tobramycin (n=10) | 1.0
  clarithromycin (n=9) | 0.9
  moxifloxacin (n=9) | 0.9
  aciclovir (n=7) | 0.7
  clindamycin (n=7) | 0.7
  other beta-lactam antibacterials (n=5) | 0.5
  ampicillin (n=4) | 0.4
  fosfomycin (n=4) | 0.4
  linezolid (n=4) | 0.4
  amikacin (n=3) | 0.3
  amphotericin B (n=3) | 0.3
  bactrim (n=3) | 0.3
  flucloxacillin (n=3) | 0.3
  rifampicin (n=3) | 0.3
  unacid (n=3) | 0.3
  benzylpenicillin (n=2) | 0.2
  beta-lactam antibacterials, penicillins (n=2) | 0.2
  ceftriaxone (n=2) | 0.2
  colistin (n=2) | 0.2
  doxycycline (n=2) | 0.2
  ganciclovir (n=2) | 0.2
  tazobactam (n=2) | 0.2
  amoxi-clavulanico (n=1) | 0.1
  antibiotics (n=1) | 0.1
  azithromycin (n=1) | 0.1
  cefotaxime (n=1) | 0.1
  cefuroxime (n=1) | 0.1
  chloramphenicol (n=1) | 0.1
  clemizole penicillin (n=1) | 0.1
  penicillin not otherwise specified (n=1) | 0.1
  piperacillin with tazobactam (n=1) | 0.1
  teicoplanin (n=1) | 0.1
  tienam (n=1) | 0.1

10. Secondary Outcome: Change of Antibiotic Treatment From Tygacil to Alternative Antibiotic
Description: Reasons for change in antibiotic treatment from Tygacil to another antibiotic.
Time Frame: Baseline to End of Treatment (up to Day 47)
Population: All participants; N = number of participants with a documented therapy switch in antibiotic treatment from Tygacil to another antibiotic; n = number of participants with specified reason for switch in antibiotic treatment . Multiple specifications were possible.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 191
percentage of participants
  Other (de-escalation) (n=80) | 7.8
  No clinical response (n=71) | 6.9
  Microbiological resistance (n=26) | 2.5
  Oral treatment continuation (n=14) | 1.4
  Intolerability (n=5) | 0.5

11. Secondary Outcome: Reasons for Utilization of Tygacil
Time Frame: Baseline to End of Treatment (up to Day 47)
Population: All participants; n = number of participants with specified reason for utilization of Tygacil.
Measure: Number; unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 1025
percentage of participants
  Failure on previous antibiotic treatment (n=549) | 53.6
  Suspicion of resistant pathogens (n=470) | 45.9
  Broad efficacy spectrum (n=463) | 45.2
  Primary (n=114) | 11.1
  Intolerability to previous antibiotic (n=21) | 2.0

12. Secondary Outcome: Overall Mortality: All Participants
Description: Deaths for any reasons occurring during the study observation period.
Time Frame: Baseline to End of Treatment (up to Day 47)
Population: All participants. Overall mortality was not calculated separately for nosocomial and community-acquired infections.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tygacil
Number analyzed (Participants) | 1025
percentage of participants | 20.0 [17.6 to 22.6]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tygacil
Serious Adverse Events (participants affected / at risk) | 245/1025
Other Adverse Events (participants affected / at risk) | 155/1025
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil (N=1025)
Multi-organ failure (General disorders) | 105
Condition aggravated (General disorders) | 47
Drug ineffective (General disorders) | 22
Concomitant disease progression (General disorders) | 11
Disease progression (General disorders) | 6
General physical health deterioration (General disorders) | 3
Death (General disorders) | 2
Brain death (General disorders) | 1
Disease recurrence (General disorders) | 1
Drug resistance (General disorders) | 1
Pyrexia (General disorders) | 1
Sepsis (Infections and infestations) | 70
Septic shock (Infections and infestations) | 35
Pneumonia (Infections and infestations) | 9
Candida sepsis (Infections and infestations) | 6
Pseudomonal sepsis (Infections and infestations) | 3
Pseudomonas infection (Infections and infestations) | 3
Aspergillosis (Infections and infestations) | 2
Catheter related infection (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 2
Fungal sepsis (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Catheter sepsis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Endocarditis staphylococcal (Infections and infestations) | 1
Enterobacter infection (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Fusarium infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Pathogen resistance (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Septic embolus (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection fungal (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac failure (Cardiac disorders) | 10
Cardiac arrest (Cardiac disorders) | 8
Myocardial infarction (Cardiac disorders) | 5
Arrhythmia (Cardiac disorders) | 3
Left ventricular failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Peritonitis (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Intestinal infarction (Gastrointestinal disorders) | 2
Pancreatitis necrotising (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Short-bowel syndrome (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 14
Cholangitis (Hepatobiliary disorders) | 2
Acute hepatic failure (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Renal failure (Renal and urinary disorders) | 13
Renal failure acute (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Blood bilirubin increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 3
C-reactive protein increased (Investigations) | 3
White blood cell count increased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Transaminases increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Ammonia increased (Investigations) | 1
Antithrombin III decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Procalcitonin increased (Investigations) | 1
Circulatory collapse (Vascular disorders) | 4
Cardiovascular insufficiency (Vascular disorders) | 3
Shock (Vascular disorders) | 3
Haemorrhage (Vascular disorders) | 2
Shock haemorrhagic (Vascular disorders) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 2
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Anastomotic complication (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Hypoxic encephalopathy (Nervous system disorders) | 2
Hypoxic encephalopathy (Nervous system disorders) | 1
Brain stem ischaemia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Coagulopathy (Blood and lymphatic system disorders) | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1
Laparotomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil (N=1025)
Drug ineffective (General disorders) | 56
Pyrexia (General disorders) | 7
Condition aggravated (General disorders) | 5
Chills (General disorders) | 1
Disease progression (General disorders) | 1
Drug effect decreased (General disorders) | 1
Drug resistance (General disorders) | 1
General physical health deterioration (General disorders) | 1
Impaired healing (General disorders) | 1
Inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema due to cardiac disease (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pathogen resistance (Infections and infestations) | 14
Infection (Infections and infestations) | 4
Candidiasis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 2
Stenotrophomonas infection (Infections and infestations) | 2
Bacterial disease carrier (Infections and infestations) | 1
Candida pneumonia (Infections and infestations) | 1
Catheter sepsis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Intestinal fistula infection (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Morganella infection (Infections and infestations) | 1
Peritoneal candidiasis (Infections and infestations) | 1
Pneumonia escherichia (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Proteus infection (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Splenic abscess (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 4
Prothrombin time prolonged (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
C-reactive protein increased (Investigations) | 3
Blood urea increased (Investigations) | 2
Lipase increased (Investigations) | 2
Transaminases increased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Clostridium difficile toxin test positive (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Interleukin level increased (Investigations) | 1
Platelet count increased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Thrombocythaemia (Blood and lymphatic system disorders) | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Glomerulonephritis (Renal and urinary disorders) | 1
Nephritis interstitial (Renal and urinary disorders) | 1
Vesical fistula (Renal and urinary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1
Somnolence (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.